CLINICAL TRIAL: NCT05575362
Title: Comparison of Epley Maneuver and COW Thorne Cooksey Exercise With Half Somersault Maneuver in Patients of BPPV
Brief Title: Comparison of Epley Maneuver and COW Thorne Cooksey Exercise With Half Somersault Maneuver in BPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zarlish
Record Dates: First submitted 2022-07-24; First posted 2022-10-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: BPPV

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epley Manuver group (Experimental): Group A is Experimental group will receive Epley's maneuver and Cawthorne Cooksey exercise for two weeks.
  Interventions: Other: Group A
- half somersault group (Active Comparator): Group B is Control group will receive Half somersault maneuver and Cawthorne Cooksey exercise for two weeks.
  Interventions: Other: Group B

INTERVENTIONS:
Other: Group A — Group A will receive Epleys maneuver and Cawthorne Cooksey exercise for two weeks.
  Arms: Epley Manuver group
Other: Group B — Group B will receive Half Somersault maneuver along with Cawthorne Cooksey exercise for two weeks.
  Arms: half somersault group

SUMMARY:
Benign paroxysmal positional vertigo is a most common cause of peripheral vestibular pathology. BPPV may be characterized by sudden changes in the position of the head, such as lying down on one or both sides, looking right or left side .it can occurs either due to canalithiasis or cupulolithiasis, displacement of otoconia or calcium carbonate crystal into fluid filled semicircular canal which sends false signals to central nervous system causing nystagmus and vertigo. BPPV is a self limiting condition characterized by episodic vertigo and nystagmus of brief duration which resolves spontaneously.

DETAILED DESCRIPTION:
BPPV is treated using canalith repositioning procedures, the most common of which is the Epley's maneuver (EM), half somersault exercises, Brandt Daroff exercise, Semont maneuver, vestibular habituation exercises, balance and eye exercises. In addition to the maneuvers, simple daily program Caw Thorne -Cooksey exercise were instructed to perform by participants to ensure clearance of the otoconia and facilitate full resolution of vertigo symptoms. These vestibular exercises involve eye, head and body movements in different directions to provoke vestibular system. It promote recovery and reduce symptoms of dizziness, unsteadiness , balance impairment and improves activity of daily living. The Otolaryngologist Caw Thorne and Cooksey develops this exercise programme in order to rehabilitate the soldier with chronic dizzeness and brain trauma. A study concluded by Ramanathan et al 2019 that Caw Thorne -Cooksey habituation exercises along with Brandt-Daroff exercises is more effective in treatment of vertigo among posterior canal BPPV subject . Caw Thorne and Cooksey exercise improves balance in old age individuals. Caw Thorne and Cooksey exercise are habituation exercise. These movements provoke patients symptoms and patients repeat these exercises until unless they no longer respond to adverse effects of these exercises .

ELIGIBILITY:
Inclusion Criteria:

* • Patients with Posterior canal BPPV.

  * Patients with recurrent episodes of vertigo for 3 months.
  * Age group 35-65years.
  * Dix-Hall-pike test positive.
  * Both gender

Exclusion Criteria:

* • Migraine related dizziness and Anxiety disorder

  * Dix hallpike test negetive
  * Other vestibular conditions are: Acoustic neuroma, Labyrinthitis, Vestibular hypofunction, Meniere's disease.
  * Any cervical pathology,
  * Visual impairment,
  * CNS Pathology:causing dizziness and vertigo
  * Other pathologies which may affect balance

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | Change from baseline, to 3rd session, 6th session and after 1 month
  The DHI is a 25-item self-report questionnaire that quantifies the impact of dizziness on daily life by measuring self-perceived handicap. Item scores are summed. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) and a minimum score of 0
vestibular activity participation scale | Change from baseline, to 3rd session, 6th session and after 1 month
  The Vestibular Activities and Participation Measure (VAP) is a 34-item self-report questionnaire that asks the individual to evaluate the effect of dizziness and/or balance problems on their ability to perform activity and participation tasks.

SECONDARY OUTCOMES:
Berg balance scale | Change from baseline, to 3rd session, 6th session and after 1 month
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MS, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Misbah, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen CC, Cho HS, Lee HH, Hu CJ. Efficacy of Repositioning Therapy in Patients With Benign Paroxysmal Positional Vertigo and Preexisting Central Neurologic Disorders. Front Neurol. 2018 Jun 29;9:486. doi: 10.3389/fneur.2018.00486. eCollection 2018. PMID 30013505
- [Background] Desai DS, Chauhan AS, Trivedi MN. Role of modified Epley's maneuver and Brandt-Daroff exercises in treatment of posterior canal BPPV: a comparative study. Int J Physiother Res. 2015;3(3):1059-64.